CLINICAL TRIAL: NCT06741007
Title: Correlation of Pelvic Sentinel Lymph Node with Superficial Vein
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Albayrak, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2828083
Record Dates: First submitted 2024-12-15; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-08

CONDITIONS: Sentinel Lymph Node; Superficial Uterine Vein; Deep Uterine Vein
Keywords: sentinel lymph node; uterine vein; uterine artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm study using ICG as a sentinel lymph node agent in early stage endometrium cancer (Experimental): Single arm study using ICG as a sentinel lymph node agent to detect the location of SLN in correlation with the presence or absence of superficial or deep uterine vein in early stage endometrial cancer
  Interventions: Procedure: Retroperitoneal pelvic lymphatic and uterine vessel dissection

INTERVENTIONS:
Procedure: Retroperitoneal pelvic lymphatic and uterine vessel dissection — ICG injection to cervix uteri at 3 and 9 o'clock followed by laparoscopic dissection of retroperitoneal space to detect uterine vessels (uterine arteries, SUVs and DUVs) bilaterally in addition to detect the location and biopsy of SLN stained by ICG.

SUMMARY:
Pelvic Sentinel Lymph Node (SLN) biopsy is an important integral part of endometrial surgery. Although SLN is usually found on internal iliac artery, location is variable. Lymphatic pathways in pelvis determines the location (Obturator, internal iliac or external iliac vessel locations). Since it is accepted that the lymphatic channel formation during embryologic life follows venous system formation investigators hypothesized that the presence or absence of superior or deep uterine vein may determine the location of sentinel lymph node

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic cancer. Treatment and prognosis depends on the surgical staging of the apparently early stage disease including the evaluation of lymphatic status of the disease. Detection of positive lymph node upstages the apparently early stage endometrial cancer. However, systematic lymphadenectomy carries immediate and long term risks for patients including bleeding, massive transfusions, prolongation of operation time, serious major vessel and major abdominal organ injury and death.

Sentinel lymph node biopsy (SLNB) procedure is the biopsy of one or two lymph node(s) which represents the lymph node basin draining the area of malignancy. This biopsy may potentially eliminate the need systemic pelvic / para-aortic lymphadenectomy which harbours potential complications. Although SLNB became an standard procedure in endometrial cancer, available data on the SLNB in endometrial cancer is variable. The relevant literature suggests that the detection rate of sentinel lymph node using various tracer agents are between %70-98, even with lower for bilateral pelvic detection and para-aortic sentinel lymph node(s). The most commonly used tracer agent is fluorescent indocyanine green (ICG). Although SLN is usually found on internal iliac artery during surgery, location is variable. Lymphatic pathways in pelvis determines the location (Obturator, internal iliac or external iliac locations). Since it is accepted that the lymphatic channel formation during embryologic life follows venous system formation investigators hypothesized that the presence or absence of right or left superior (SUV) or deep uterine vein (DUV), which actually are highly variable, may determine the location of sentinel lymph node.

So investigators aims to find any correlation between the location of SLN (obturator, external iliac and internal iliac) and the presence of SUV or DUV unilaterally or bilaterally.

ELIGIBILITY:
Inclusion Criteria:

* all women with early stage endometrial cancer who will be operated for staging

Exclusion Criteria:

Previous radiotheraphy Previous pelvic retropelvic LN dissection Women with any disease that precludes pelvic retropelvic LN dissection (such as peritoneal dialysis)

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-12-22 (Estimated); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Detection rate and localisation of SLN in correlation with the presence or absence of uterine veins bilaterally | Two years
  The location of SLN ( obturator, external iliac and internal iliac) will be defined in percentages for each side of pelvis in relation to presence or absence of uterine vessels.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ribatti D. Historical overview of lymphangiogenesis. Curr Opin Immunol. 2018 Aug;53:161-166. doi: 10.1016/j.coi.2018.04.027. Epub 2018 May 19. PMID 29787938
- [Background] Kimmig R, Thangarajah F, Buderath P. Sentinel Lymph node detection in endometrial cancer - Anatomical and scientific facts. Best Pract Res Clin Obstet Gynaecol. 2024 Jun;94:102483. doi: 10.1016/j.bpobgyn.2024.102483. Epub 2024 Feb 15. PMID 38401483